CLINICAL TRIAL: NCT01630109
Title: Metoclopramide As An Adjunct To Small Bowel Capsule Endoscopy: Rate of Complete Evaluation And Affect on Transit Times
Brief Title: Study of Metoclopramide in Small Bowel Capsule Endoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Steven Brooks, DO/Internal Medicine Resident, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GRMC120006
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Pill Capsule Endoscopy Completion Rates
MeSH Terms: interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Metoclopramide 5 mg (Active Comparator): Pro-motility agent
  Interventions: Drug: Metoclopramide
- Metoclopramide 10 mg (Active Comparator): Pro-motility agent
  Interventions: Drug: Metoclopramide
- Placebo control (Placebo Comparator): Placebo to be used as the control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoclopramide — A one time dose of either Metoclopramide 5 mg or 10 mg (or placebo) given orally 30 minutes prior to pill capsule endoscopy.
  Other Names: Brand name of Metoclopramide is Reglan
  Arms: Metoclopramide 10 mg; Metoclopramide 5 mg
Drug: Placebo — A placebo capsule made to look like the metoclopramide capsule.
  Arms: Placebo control

SUMMARY:
Patients undergoing small bowel capsule endoscopy will be randomized into 3 study groups to either receive 5 mg of metoclopramide, 10 mg of metoclopramide, or a placebo 30 minutes prior to swallowing the Pill Cam. This is a randomized, double-blind, placebo-controlled design. The outcomes to be assessed are capsule study completion rates, gastric transit time, small bowel transit time, and the effect of diabetes on pill capsule completion rates. The purpose of the study is to assess if metoclopramide given prior to pill capsule endoscopy has any effect on pill capsule completion rate, gastric transit time, small bowel transit time, and pill capsule completion rates in diabetes.

DETAILED DESCRIPTION:
Pill Capsule Endoscopy allows Gastroenterologists to visualize the mucosa of the small bowel beyond the reach of any endoscope and to an extent never before possible. It involves the ingestion of a small pill camera approximately the size of a large vitamin. 8 hours of images are transmitted to a sensor worn around the patient's waist. At the conclusion of the test, these images are downloaded to a computer for physician review. Meanwhile, the PillCam™ passes naturally through the digestive system and does not require retrieval.

Many of these pill capsule studies are incomplete due to failure of the pill capsule to reach the colon. Metoclopramide (brand name Reglan) is an anti-emetic that also has known pro-motility effects in the GI tract. The thought behind this study is that metoclopramide will increase the rate of passage of the pill capsule through the GI tract allowing a higher completion rate of the pill capsule studies.

Patients scheduled for pill capsule endoscopy will be approached on the morning of their procedure to inform them of the research study. After proper consent is obtained the patient will receive either 5 mg Metoclopramide, 10 mg Metoclopramide, or a placebo pill 30 minutes prior to their pill capsule study. The pill capsule camera records 8 hours worth of data. The patient will return at the conclusion of their study to turn in their recorder. The ordering gastroenterologist will then read the study. Information regarding pill capsule completion (pill capsule goes through the ileocecal valve), gastric transit time, and small bowel transit time will then be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18 undergoing pill capsule endoscopy to investigate unexplained rectal bleeding, anemia, iron deficiency, abdominal pain, altered bowel habits, and/or weight loss.

Exclusion Criteria:

* Inability to sign consent for research participation
* Inability to swallow PillCam™, placebo, or metoclopramide capsule
* Known hypersensitivity/allergy to metoclopramide
* Active congestive heart failure or respiratory failure requiring ventilator assistance
* Presence of cardiac pacemaker or implanted electromedical device
* Known bowel obstruction/stricture/fistula or intrauterine pregnancy
* Known history of Whipple procedure (pancreaticoduodenectomy), Billroth II surgery (partial gastrectomy with gastrojejunostomy), or gastric bypass surgery due to risk of capsule retention in a blind intestinal limb necessitating surgical retrieval
* Known history of seizure disorder, renal failure requiring dialysis, or pheochromocytoma
* Lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven D Brooks, D.O., Principal Investigator — Ascension Health
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited from December 2012 to June 2013. The subjects were recruited in the Medical Procedures Unit at Genesys Regional Medical Center.
Pre-assignment Details: No events to report.
Period: Overall Study
Arm/Group | Metoclopramide 5 mg | Metoclopramide 10 mg | Placebo Control
Started | 1 | 1 | 3
Completed | 1 | 1 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide 5 mg | Metoclopramide 10 mg | Placebo Control | Total
Number analyzed (Participants) | 1 | 1 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 3 | 5
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (0) | 59 (0) | 46 (12.76) | 50.20 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2
  Male | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Difference in Treatment vs. Placebo in Pill Capsule Completion Rates
Description: This study is investigating whether there is a difference in pill capsule completion rates between a treatment group (metoclopramide) vs. placebo. It is also looking at differences in completion rates between two different doses of metoclopramide (5 mg vs. 10 mg).
Time Frame: 12 hours
Measure: Number; unit: percentage of complete capsule studies
Arm/Group | Metoclopramide 5 mg | Metoclopramide 10 mg | Placebo Control
Number analyzed (Participants) | 1 | 1 | 3
percentage of complete capsule studies | 100 | 0 | 100

2. Secondary Outcome: Differences in Gastric Transit Time in Treatment vs. Placebo in Pill Capsule Studies
Description: This study will investigate whether treatment with metoclopramide (5 mg or 10 mg) vs. placebo will affect gastric transit time.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Metoclopramide 5 mg | Metoclopramide 10 mg | Placebo Control
Number analyzed (Participants) | 1 | 1 | 3
minutes | 15 (0) | 57 (0) | 88 (106.12)

3. Secondary Outcome: Differences in Small Bowel Transit Time in Treatment vs. Placebo in Pill Capsule Studies
Description: This study will investigate whether there is a difference in small bowel transit time in pill capsule studies with treatment with metoclopramide (5 mg or 10 mg) vs. placebo.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Metoclopramide 5 mg | Metoclopramide 10 mg | Placebo Control
Number analyzed (Participants) | 1 | 1 | 3
minutes | 53 (0) | 218 (0) | 301 (114.45)

4. Secondary Outcome: Difference in Pill Capsule Completion Rates in Diabetics vs. Non-diabetics
Description: This study will investigate whether there is any difference in pill capsule completion rates in patients who are diabetic vs. those who are not diabetic.
Time Frame: 12 hours
Measure: Number; unit: Percentage of complete studies
Groups:
- Metoclopramide 5 mg (Diabetics); Metoclopramide 10 mg (Diabetics): Pro-motility agent given to diabetic patients
- Placebo Control (Diabetics): Placebo to be used as the control group in diabetic patients
- Metoclopramide 5 mg (Non-diabetic); Metoclopramide 10 mg (Non-diabetic): Pro-motility agent given to non-diabetic patients
- Placebo (Non-diabetic): Placebo control given to non-diabetics
Arm/Group | Metoclopramide 5 mg (Diabetics) | Metoclopramide 10 mg (Diabetics) | Placebo Control (Diabetics) | Metoclopramide 5 mg (Non-diabetic) | Metoclopramide 10 mg (Non-diabetic) | Placebo (Non-diabetic)
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 2
Percentage of complete studies |  |  | 100 | 100 | 0 | 100

ADVERSE EVENTS:
Arm/Group | Metoclopramide 5 mg | Metoclopramide 10 mg | Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/3

LIMITATIONS AND CAVEATS:
The main limitation of this study was that there was a lower number of capsule studies performed at the study center than anticipated so it was difficult to find patients to enroll.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No